CLINICAL TRIAL: NCT00772252
Title: Oxidative Stress and Microcirculation in Patient With Hepatic Failure Undergoing Liver Support Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yu-Chang Yeh / Doctor, NTUH
Other Study IDs: 200806004R
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Liver Failure; Critical Care
Keywords: Liver support treatment
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patient with hepatic failure undergoing liver support treatment in surgical intensive care unit
  Interventions: Other: liver support treatment

INTERVENTIONS:
Other: liver support treatment — plasma exchange for liver support treatment

SUMMARY:
Background: In patients undergoing hemodialysis or hemofiltration will suffer from the injury of reactive oxidative species. Oxidative stress will affect cell membrane, protein, and DNA. It will damage the cell and result in organ dysfunction. We believe that in patients, who have acute hepatic failure, undergoing plasma exchange or Molecular Absorbent Recirculating System for bridge therapy will suffer from the injury of reactive oxidative species, too. It will damage the kidney, lung, cerebral cortex, and other organs. It may result in death before the recovery of liver function or undergoing liver transplantation.

Aims: 1. Investigate the severity of oxidative stress and risk factors of high oxidative stress in acute hepatic failure patient undergoing plasma exchange or Molecular Absorbent Recirculating System. 2. Investigate the microcirculation status and risk factors in acute hepatic failure patient undergoing plasma exchange or Molecular Absorbent Recirculating System. 3. Study the relationship between oxidative stress and microcirculation status. 4. Study the correlation between oxidative stress and prognosis. 5. Study the correlation between microcirculation status and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Patients with acute deterioration on Chronic liver failure, who required liver support treamtment
3. Patients with acute liver failure due to acute hepatitis, who reauired liver support treatment
4. Patients with acute liver dysfunction within 7 days after liver transplantation, who required liver support treatment

Exclusion Criteria:

1. Age > 70 years old
2. Cancer, not curable
3. Patients who had used of antioxidant therapy within 24 hours before study
4. Patients who had received hyperbaric oxygen therapy within 24 hours before study
5. Patients who had received peroxide treatment within 24 hours before study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients require liver support treatment
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, Bacehlor, Study Director — Department of Anesthesiology, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan